CLINICAL TRIAL: NCT04194632
Title: Right Ventricular Pacing to Treat Right Ventricular Failure: A Single Arm Hemodynamic Study
Brief Title: Right Ventricular Pacing in Pulmonary Arterial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-25983
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Artery Hypertension; Right Ventricular Dysfunction
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Ventricular Dysfunction, Right

STUDY DESIGN:
Intervention Model Description: As described previously, patients will undergo measurements at baseline, with pacing, and post pacing and will thus function as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All patients will undergo hemodynamic measurements at baseline, with the intervention, and post-intervention thus serving as their own control.
  Interventions: Procedure: Temporary right ventricular pacing

INTERVENTIONS:
Procedure: Temporary right ventricular pacing — As described previously. Patients will undergo temporary pacing at the site of latest endocardial activation with measurement of hemodynamic effects.

SUMMARY:
In pulmonary arterial hypertension (PAH), progressive pulmonary vascular remodeling leads to supraphysiologic right ventricular (RV) afterload. Pharmacologic trials have shown that aggressive upfront treatment reversing pulmonary vascular remodeling successfully increases RV function and improves survival. To date, however, there are no proven treatments that target RV contractile function.

Echocardiographic studies of RV dysfunction in the setting of pressure overload have demonstrated intra and interventricular dyssynchrony even in the absence of overt right bundle branch block (RBBB).

Electrophysiologic studies of patients with chronic thromboembolic disease (CTEPH) at the time of pulmonary endarterectomy have shown prolongation of action potential and slowed conduction in the right ventricle which has correlated with echocardiographic measures of dyssynchrony.

Cardiac MRI measures of RV strain in patients with PAH demonstrated simultaneous initiation of RV and left ventricular (LV) contraction, but delayed peak RV strain suggesting that interventricular dyssynchrony is a mechanical rather than electrical phenomenon.

Prior studies of RV dysfunction in an animal model, computer model, congenital heart disease, and CTEPH have suggested acute hemodynamic benefits of RV pacing. However, RV pacing has not been studied in patients with PAH. Furthermore, it remains unclear if pacing particular regions of the RV can achieve a hemodynamic benefit and what cost this hemodynamic improvement may incur with regards to myocardial energetics and wall stress.

Therefore, the investigators propose to examine RV electrical activation in PAH, map the area of latest activation, and then evaluate the hemodynamic and energetic effects of RV pacing in these patients.

DETAILED DESCRIPTION:
Research procedures in chronological order:

1. Baseline clinical variables will be prospectively determined and then obtained retrospectively from the clinical assessment of individual pulmonary hypertension team physicians via chart review. The most recent transthoracic echocardiogram will also be evaluated and routine clinical variables including tricuspid annular plane systolic excursion (TAPSE), RV fractional area change (FAC), RV outflow tract (OT) and LVOT velocity time integral (VTI), and ejection fraction (EF) will be extracted.
2. All patients will have cardiac MRI performed prior to the procedure to allow precise measurement of right ventricular volumes as well as LV volumes, RVEF, and LVEF. Gadolinium enhancement using gadolinium contrast will be measured.
3. Standard of care right heart catheterization (RHC) will be performed on the day of the research procedure.
4. Radial arterial pressure will be used for periprocedural monitoring as well as for sampling of arterial oxygen content and arterial oxygen lactate.
5. Myocardial energetics will be assessed via sampling of coronary sinus venous blood with measurement of oxygen saturation and lactate.
6. Following the standard of care RHC, endocardial mapping will be performed. After pressure-volume measurements are obtained (step 7), pacing will be performed from the right atrium (RA), His bundle, and RV at the site of the latest activation with repeat measurements of pressure-volume relationships.
7. Once endocardial mapping is complete, a 7-French Millar conductance catheter will be placed into the RV and used to obtain pressure-volume data for the RV using the INCA PV signal processor. The Valsalva maneuver will be used to generate a series of PV-loops reflecting preload reduction subsequently allowing for the calculation of a load independent measure of contractility, the end systolic pressure volume relationship (Ees). RV afterload will be measured as effective arterial elastance (Ea) and V-A coupling will be assessed by the ratio of Ees/Ea. Myocardial energetics will be assessed via PV area (PVA) and calculation of the transmyocardial arteriovenous oxygen extraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for a clinically indicated right heart catheterization to either diagnose pulmonary arterial hypertension prior to initiating therapies or monitor response to ongoing therapies in patients with diagnosed pulmonary arterial hypertension.
* Patients with pulmonary arterial hypertension with or without significant right ventricular dysfunction as assessed by baseline echocardiography and standard of care right heart catheterization
* Functional class 2 or 3 symptoms
* Are able to undergo cardiac MRI, endocardial mapping, and pressure volume measurements
* English speaking
* All patients will be required to have evidence of right ventricular hypertrophy or conduction delay (QRS > 130ms) on surface ECG

Exclusion Criteria:

* Preexisting left bundle branch block, current atrial fibrillation, or pacemaker/ defibrillators
* Functional class 4 symptoms
* Patients treated with parenteral or subcutaneous therapies for pulmonary hypertension
* Contraindication to right heart catheterization including significant thrombocytopenia (platelets < 50,000), coagulopathy (INR > 1.8), or pregnancy as determined by routine screening laboratory work
* Mean pulmonary artery pressure less than 25 mmHg as determined by the right heart catheterization on the day of the study procedure
* Pulmonary capillary wedge pressure greater than or equal to 15 mmHg as determined by the right heart catheterization on the day of the study procedure
* Severe tricuspid regurgitation as determined by baseline transthoracic echocardiogram.
* Left ventricular dysfunction (EF < 50%) as determined by baseline transthoracic echocardiogram.
* Inability to complete cardiac MRI or transthoracic echocardiography
* Patients with confounding systemic disease specifically portopulmonary hypertension and scleroderma associated pulmonary hypertension
* Patients otherwise deemed not appropriate for the study as determined by the study investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-05 (Estimated); Study Completion 2021-12-05 (Estimated)

PRIMARY OUTCOMES:
Change in contractility (Ees) | During procedure. The measurement will be taken pre-RV pacing, with RV pacing, and 5 minutes after RV pacing. All catheters will then be removed and the study will be completed.
  This is an invasive measure of the contractile strength of the right ventricle that is measured using pressure volume measurements from within the ventricle itself.

SECONDARY OUTCOMES:
Change in stroke volume | During procedure. The measurement will be taken pre-RV pacing, with RV pacing, and 5 minutes after RV pacing. All catheters will then be removed and the study will be completed.
  This is an invasive measure of the amount of blood ejected by the heart with each heart beat.
Pressure-volume loop area | During procedure. The measurement will be taken pre-RV pacing, with RV pacing, and 5 minutes after RV pacing. All catheters will then be removed and the study will be completed.
  The pressure-volume loop area will be calculated to assess right ventricular myocardial oxygen consumption
Coronary sinus oxygen saturation | During procedure. The measurement will be taken pre-RV pacing, with RV pacing, and 5 minutes after RV pacing. All catheters will then be removed and the study will be completed.
  Global myocardial oxygen consumption will also be assessed via measurement of the coronary sinus oxygen saturation.

CONTACTS AND LOCATIONS:
Overall Officials: Liviu Klein, MD, Principal Investigator — University of California, San Francisco; Benjamin W Kelemen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalogeropoulos AP, Georgiopoulou VV, Howell S, Pernetz MA, Fisher MR, Lerakis S, Martin RP. Evaluation of right intraventricular dyssynchrony by two-dimensional strain echocardiography in patients with pulmonary arterial hypertension. J Am Soc Echocardiogr. 2008 Sep;21(9):1028-34. doi: 10.1016/j.echo.2008.05.005. Epub 2008 Jun 16. PMID 18558476
- [Background] Hardziyenka M, Campian ME, Bouma BJ, Linnenbank AC, de Bruin-Bon HA, Kloek JJ, van der Wal AC, Baan J Jr, de Beaumont EM, Reesink HJ, de Bakker JM, Bresser P, Tan HL. Right-to-left ventricular diastolic delay in chronic thromboembolic pulmonary hypertension is associated with activation delay and action potential prolongation in right ventricle. Circ Arrhythm Electrophysiol. 2009 Oct;2(5):555-61. doi: 10.1161/CIRCEP.109.856021. Epub 2009 Aug 4. PMID 19843924
- [Background] Marcus JT, Gan CT, Zwanenburg JJ, Boonstra A, Allaart CP, Gotte MJ, Vonk-Noordegraaf A. Interventricular mechanical asynchrony in pulmonary arterial hypertension: left-to-right delay in peak shortening is related to right ventricular overload and left ventricular underfilling. J Am Coll Cardiol. 2008 Feb 19;51(7):750-7. doi: 10.1016/j.jacc.2007.10.041. PMID 18279740
- [Background] Hardziyenka M, Surie S, de Groot JR, de Bruin-Bon HA, Knops RE, Remmelink M, Yong ZY, Baan J Jr, Bouma BJ, Bresser P, Tan HL. Right ventricular pacing improves haemodynamics in right ventricular failure from pressure overload: an open observational proof-of-principle study in patients with chronic thromboembolic pulmonary hypertension. Europace. 2011 Dec;13(12):1753-9. doi: 10.1093/europace/eur189. Epub 2011 Jul 21. PMID 21784747
- [Background] Handoko ML, Lamberts RR, Redout EM, de Man FS, Boer C, Simonides WS, Paulus WJ, Westerhof N, Allaart CP, Vonk-Noordegraaf A. Right ventricular pacing improves right heart function in experimental pulmonary arterial hypertension: a study in the isolated heart. Am J Physiol Heart Circ Physiol. 2009 Nov;297(5):H1752-9. doi: 10.1152/ajpheart.00555.2009. Epub 2009 Sep 4. PMID 19734361
- [Background] Lumens J, Arts T, Broers B, Boomars KA, van Paassen P, Prinzen FW, Delhaas T. Right ventricular free wall pacing improves cardiac pump function in severe pulmonary arterial hypertension: a computer simulation analysis. Am J Physiol Heart Circ Physiol. 2009 Dec;297(6):H2196-205. doi: 10.1152/ajpheart.00870.2009. Epub 2009 Oct 16. PMID 19837949
- [Background] Janousek J, Kovanda J, Lozek M, Tomek V, Vojtovic P, Gebauer R, Kubus P, Krejcir M, Lumens J, Delhaas T, Prinzen F. Pulmonary Right Ventricular Resynchronization in Congenital Heart Disease: Acute Improvement in Right Ventricular Mechanics and Contraction Efficiency. Circ Cardiovasc Imaging. 2017 Sep;10(9):e006424. doi: 10.1161/CIRCIMAGING.117.006424. PMID 28877886